CLINICAL TRIAL: NCT01330797
Title: The Effect of Ranibizumab on Eye Lens Opacity in Cases With Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Mehmet Baykara, MD, Uludag University School of Medicine
Other Study IDs: GOZ-1
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-01

CONDITIONS: Age-Related Macular Degeneration; Cataract
Keywords: Cataract; Intravitreal; Ranibizumab; LOCS III
MeSH Terms: conditions — Macular Degeneration; Cataract

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LOCS III: Cohort is composed of cases with a diagnosis of wet age-related macular degeneration and those that received intravitreal ranibizumab

SUMMARY:
Purpose To evaluate the cataractogenic effect of intravitreal ranibizumab with the use of Lens Opacity Classification System III (LOCS III).

Settings Cases with a diagnosis of wet AMD were included in this university practice based prospective study.

Methods All cases had monthly injections of intravitreal ranibizumab in the first 3 months; subsequently an OCT-guided pro re nata injection regimen has been adopted. All cases had a comprehensive eye examination and LOCS III evaluation at baseline and 1, 3, 6 and 12 months after the initial injection. Examination outcomes and change from baseline in LOCS III grades at 12 months were recorded.

Results Eighteen eyes of 13 cases (7 female, 6 male) were included in this study. The mean age at the baseline was 75,3 + 6,6 years. A mean of 3,4 + 0,7 injections were given on each eye. Mean follow-up was 13,83 + 2,33 months. Baseline mean visual acuity improved from 1,04 + 0,10 logMAR units to 0,76 + 0,26 logMAR units after 3 injections (P < 0.05). At the 12th month of follow-up mean visual acuity was 0,71 + 0,27 logMAR units. According to LOCS III grades none of the cases had a prominent change in nuclear color, nuclear opalescence, cortical and posterior subcapsular opacification throughout the follow-up. IOP remained stable at all follow-up points. No complications were recorded throughout the study.

Conclusion Intravitreal ranibizumab is an efficient treatment in wet AMD. Results of LOCS III assessments in this pilot study suggest that intravitreal ranibizumab has no effect on the progression of lens opacity.

DETAILED DESCRIPTION:
In the last decade, significant progress has been made in the treatment of wet AMD. At the present intravitreal anti-VEGF therapy has become the mainstay of treatment. Nevertheless, intravitreal application is a hazardous procedure with a wide range of complications. Endophthalmitis, intraocular pressure (IOP) elevation, retinal detachment, vitreous hemorrhage, and cataract are among the major complications.

The current study is focused on the cataractogenic potential of intravitreal ranibizumab. Cataract formation following intravitreal application is frequently associated with an inadvertent trauma at the procedure. However, occasionally the drug -itself- may precipitate cataract formation. Accelerated formation of cataract, has previously been shown as a possible cause of decreased visual acuity, in some cases who received intravitreal injections of triamcinolone. However, no prospective study has, as yet, assessed anti-VEGF agent related cataract progression in cases of AMD. Herein, the investigators have investigated the cataractogenic effect of intravitreal ranibizumab by using the Lens Opacity Classification System III (LOCS III).

ELIGIBILITY:
Inclusion Criteria:

* Neovascular age-related macular degeneration cases undergoing ranibizumab treatment
* Phakic patients

Exclusion Criteria:

* History of previous injections of a triamcinolone or anti-VEGF drug
* Individuals that had undergone cataract extraction
* Cases that had other intraocular surgery within the last 3 months
* Cases that had any laser treatment within 1 month (including YAG laser iridotomy)
* Cases that are using systemic steroids or anti-glaucomatous drops

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neovascular age-related macular degeneration cases undergoing ranibizumab treatment
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Lens Opacity Classification System (LOCS) III grades | Change from baseline in LOCS III grades at 12 months are recorded.
  Evaluation of lens status are assessed according to LOCS III standards. Attributes of LOCS III; nuclear color (NC), nuclear opalescence (NO), cortical opacity (CO), and posterior subcapsular opacity (PSC) are graded for each eye. Each attribute range from 0.1 (clear) to 6.9 (most advanced) in 0.1 increments.Change from baseline in LOCS III grades at 1 month, 3 months, 6 months and at 12 months are recorded.

SECONDARY OUTCOMES:
Best corrected visual acuity | change from baseline in LOCS III grades at 12 months are recorded
  Best corrected visual acuity of each individual is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Baykara, M.D, Principal Investigator — Uludag University School of Medicine, Department Of Ophthalmlogy
Locations (1):
- Uludag University School of Medicine, Department of Ophthalmology, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Sampat KM, Garg SJ. Complications of intravitreal injections. Curr Opin Ophthalmol. 2010 May;21(3):178-83. doi: 10.1097/ICU.0b013e328338679a. PMID 20375895
- [Background] Jonas JB. Intravitreal triamcinolone acetonide: a change in a paradigm. Ophthalmic Res. 2006;38(4):218-45. doi: 10.1159/000093796. Epub 2006 Jun 6. PMID 16763379
- [Background] Jonas JB, Kreissig I, Degenring RF. Cataract surgery after intravitreal injection of triamcinolone acetonide. Eye (Lond). 2004 Apr;18(4):361-4. doi: 10.1038/sj.eye.6700654. PMID 15069430
- [Background] Regillo CD, Brown DM, Abraham P, Yue H, Ianchulev T, Schneider S, Shams N. Randomized, double-masked, sham-controlled trial of ranibizumab for neovascular age-related macular degeneration: PIER Study year 1. Am J Ophthalmol. 2008 Feb;145(2):239-248. doi: 10.1016/j.ajo.2007.10.004. PMID 18222192
- [Background] Chylack LT Jr, Gross GN, Pedinoff A; Ciclesonide Lenticular Safety Study Group. A randomized, controlled trial to investigate the effect of ciclesonide and beclomethasone dipropionate on eye lens opacity. J Asthma. 2008 Dec;45(10):893-902. doi: 10.1080/02770900802353636. PMID 19085579